CLINICAL TRIAL: NCT00112645
Title: A Phase I Study to Examine the Toxicity of Allogeneic Stem Cell Transplantation for Pediatric Solid Tumors With Relapsed or Therapy Refractory Disease
Brief Title: Donor Stem Cell Transplant in Treating Young Patients With Relapsed or Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: PSCI-20615; CDR0000430441 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2005-06-02; First posted 2005-06-03 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2011-02

CONDITIONS: Neuroblastoma; Sarcoma; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: unspecified childhood solid tumor, protocol specific; recurrent neuroblastoma; recurrent Ewing sarcoma/peripheral primitive neuroectodermal tumor; recurrent childhood rhabdomyosarcoma
MeSH Terms: conditions — Neuroblastoma; Sarcoma; Neuroectodermal Tumors, Primitive, Peripheral | interventions — Antilymphocyte Serum; Busulfan; Cyclosporine; Melphalan; Methotrexate; Methylprednisolone; Peripheral Blood Stem Cell Transplantation; Cord Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: anti-thymocyte globulin
Drug: busulfan
Drug: cyclosporine
Drug: melphalan
Drug: methotrexate
Drug: methylprednisolone
Procedure: allogeneic bone marrow transplantation
Procedure: peripheral blood stem cell transplantation
Procedure: umbilical cord blood transplantation

SUMMARY:
RATIONALE: A peripheral stem cell, bone marrow, or umbilical cord blood transplant may be able to replace blood-forming cells that were destroyed by chemotherapy and radiation therapy. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving busulfan and melphalan with or without antithymocyte globulin before transplant and cyclosporine with methylprednisolone or methotrexate after transplant may stop this from happening.

PURPOSE: This phase I trial is studying the side effects of donor stem cell transplant in treating young patients with relapsed or refractory solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxicity of allogeneic hematopoietic stem cell transplantation, in terms of the incidence of grade 3-4 acute graft-versus-host disease, in young patients with relapsed or refractory solid tumors.
* Determine the incidence of transplant-related mortality at 100 days post-transplantation in these patients.

OUTLINE:

* Conditioning: Patients receive busulfan IV or orally 4 times daily on days -8 to -5 (a total of 16 doses) and melphalan IV over 15-20 minutes on days -4 to -2. Patients with an unrelated donor also receive anti-thymocyte globulin IV on days -4 to -2.
* Allogeneic hematopoietic stem cell transplantation (SCT): Patients undergo allogeneic hematopoietic SCT on day 0.
* Post-transplant graft-versus-host disease (GVHD) prophylaxis: Patients who undergo cord blood SCT receive cyclosporine and methylprednisolone for graft-versus-host disease (GVHD) prophylaxis. Patients who undergo peripheral blood or bone marrow SCT receive cyclosporine and methotrexate (short course) for GVHD prophylaxis.

After completion of study treatment, patients are followed at 1, 3, 6, and 12 months and then annually thereafter.

PROJECTED ACCRUAL: A total of 10 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of relapsed or refractory solid tumor, including, but not limited to, relapsed neuroblastoma, relapsed Ewing's sarcoma, and relapsed rhabdomyosarcoma
* No isolated local disease recurrence at the site of the primary tumor > 1 year after completion of prior therapy
* No brain tumor or brain metastases
* Related or unrelated hematopoietic stem cell donor available, meeting 1 of the following criteria:

  * Matched for HLA-A, -B, -C, -DR, and -DQ (9/10 or 10/10 allelles) (marrow or peripheral blood)
  * Matched for HLA-A, -B, and -DR (5/6 or 6/6 allelles) (cord blood)

    * Cord blood specimen must contain ≥ 2 x 10 ^7 nucleated cells/kg body weight

PATIENT CHARACTERISTICS:

Age

* 30 and under

Performance status

* ECOG 0-1 OR
* Lansky 80-100%

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Bilirubin ≤ 3.0 mg/dL

Renal

* Creatinine clearance ≥ 50 mL/min

Cardiovascular

* Ejection fraction ≥ 50%

Pulmonary

* DLCO ≥ 70% OR
* O_2 saturation ≥ 95% on room air

Other

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Prior autologous stem cell transplantation allowed

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2005-04; Primary Completion 2010-04 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth G. Lucas, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Hershey Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States